CLINICAL TRIAL: NCT03272191
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Cardiovascular Effects of Autologous ADSC Implantation by a Catheter Delivery System In Patients During the Subacute Recovery Phase of ST-Elevation MI
Brief Title: Study to Assess Safety & Effects of Autologous ADSCs During Recovery Phase of ST-Elevation MI Effects of Autologous ADSC Implantation During Subacute Recovery Phase of ST-Elevation Myocardial Infarction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ME-SMI-001
Record Dates: First submitted 2013-10-28; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-07

CONDITIONS: Subacute Myocardial Infarction
Keywords: MI; Infarction; Infarct; Subacute MI; stem cell
MeSH Terms: conditions — Infarction | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Liposuction and stem cell implantation — The adipose tissue specimen will be collected mainly from the patient's abdomen using a liposuction cannula. The adipose tissue may be collected from other areas if necessary The adipose tissue is transferred to the laboratory for separation of the adipose tissue-derived stem cells, which are then transferred to an injection/infusion catheter for delivery into the akinetic myocardial scar in the region of a previous infarct

SUMMARY:
The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe? and 2) Is treatment effective in improving cardiac function and clinical outcomes?

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center study of ASC implantation using a catheter delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The injection catheter will be used for delivery of the ASCs therapy.

The adipose tissue specimen will be collected mainly from the patient's abdomen using a liposuction cannula. The adipose tissue may be collected from other areas if necessary The adipose tissue is transferred to the laboratory for separation of the adipose tissue-derived stem cells, which are then transferred to an injection/infusion catheter for delivery into the akinetic myocardial scar in the region of a previous infarct

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Defined subacute myocardial infarction between 9-90 days from screening
* Left ventricular ejection fraction at screening of ≤ 50%, with 2 or more contiguous areas of severe wall motion abnormality on resting echocardiography.
* Patients must have a minimum myocardial wall thickness of 5mm
* Need or feasibility for re-vascularization has been ruled out by coronary angiogram or noninvasive stress testing.
* Stable for at least 14 days on optimal medical management including:
* Plavix/asprin therapy, anticoagulation therapy, cholesterol lowering agent, beta blocker, ACE inhibitor or ARB blocker Up to date on all age and gender appropriate cancer screening per American Cancer Society (Refer to section 9.3 for more details).

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* NYHA CHF Class 4
* Severe valvular or other non-ischemic myocardial disease.
* Mechanical complications of the index acute myocardial infarction including but not limited to rupture of the mitral valve with resultant development of mitral regurgitation, rupture of the left ventricular free wall and rupture of the interventricular septum.
* Previous severe reaction to radiocontrast agents
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Serum creatinine > 2.5 mg/dL or end stage renal disease unless on dialysis.
* Active infectious disease and/or known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis. If the panel includes antibodies to the HBV-cAg and HBV-sAg, then an expert will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection within one week of enrollment.
* Cerebrovascular accident within 6 months prior to study entry
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Improved cardiac function | 3 and 6 months after intervention
  Improvement is observed in cardiac function as assessed by echocardiographic LV function (EF)

SECONDARY OUTCOMES:
Adverse Event | Duration of study
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States